CLINICAL TRIAL: NCT06477562
Title: The Success Rate and Associated Factors for Surveillance Endoscopy After Proximal Gastrectomy With Double Tract Reconstruction: Multicenter Retrospective Study
Brief Title: Surveillance Endoscopy After Proximal Gastriectomy With Double Tract Reconstruction.
Status: Completed | Type: Observational
Sponsor: Saint Vincent's Hospital, Korea (Other)
Responsible Party: Principal Investigator, Ki Bum Park, Doctor, Saint Vincent's Hospital, Korea
Other Study IDs: VC24WADI0021
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Gastric Cancer; Proximal Gastric Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Proximal gastrectomy with double tract reconstruction group
  Interventions: Other: Endoscopy

INTERVENTIONS:
Other: Endoscopy — surveillance endoscopy was routinely performed to the patients with proximal gastrectomy with double tract reconstruction group.

SUMMARY:
The primary purpose of surveillance endoscopy after gastric cancer surgery is to detect malignancy recurrence in the remnant stomach. This study aims to analyze the rate of proper remnant stomach observation following proximal gastrectomy(PG) with double tract reconstruction (DTR). Data from patients who underwent PG with DTR for gastric cancer at six institutions in South Korea from 2011 to 2023 were included. Clinicopathological and serial endoscopic data were retrospectively reviewed and analyzed. Successful surveillance endoscopy was defined as obtaining an endoscopic image of the pyloric antrum. Factors associated with successful endoscopy were analyzed using a mixed-effects logistic regression model. A total of 634 surveillance endoscopies were performed on 160 patients after PG with DTR. The median duration from surgery to the endoscopy was 17.5 months (range, 0-137 months). The success rate of the endoscopies was 75.6%, with a mean time of 271.7±300.5 seconds to reach the pyloric antrum. The average total procedure time for successful endoscopic examinations was 439.4±336.0 seconds, compared to 373.7±326.0 seconds for failed examinations. (p=0.033). Among patients who underwent the procedure twice or more, 6.5% had all endoscopic examinations fail, while 2.8% of those who underwent the procedure three times or more experienced failure in all examinations. Factors associated with successful endoscopy included longer procedure time (OR 1.32, 95% CI 1.01-1.72), endoscopy performed by a non-surgeon (OR 0.19, 95% CI 0.11-0.36), longer duration after surgery (OR 1.33, 95% CI 1.02-1.72) and younger age (OR 0.70, 95% CI 0.49-0.97). Understanding the anatomic alterations after PG with DTR is crucial for the success of surveillance endoscopy. Additionally, the duration from surgery to endoscopy is associated with the success of the examination, and the rate of failure across all serial endoscopies is very low. Therefore, clinicians should perform endoscopies with sufficient procedure time and conduct endoscopies regardless of the failure of previous examinations.

ELIGIBILITY:
Inclusion Criteria:

Patients who underwent proximal gastrectomy with double tract reconstruction and had at least one postoperative surveillance endoscopy.

Exclusion Criteria:

Patients who did not undergo postoperative surveillance endoscopy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent proximal gastrectomy with double tract reconstruction and had at least one postoperative surveillance endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Successful surveillance endoscopy | Routine endoscopic surveillance was performed 6 months after surgery.
  Obtaining an endoscopic image of the pyloric antrum.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiwon Seo, Suwon, Gyeong-Gi-Do, South Korea

IPD SHARING:
Plan to Share IPD: No